CLINICAL TRIAL: NCT01595360
Title: A Phase 1, Randomized, Open, Controlled, Comparative Safety, Tolerability and Efficacy Study of TT-173 in Healthy Volunteers After Tooth Extraction
Brief Title: Safety, Tolerability and Efficacy Study of TT-173 in Healthy Volunteers After Tooth Extraction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thrombotargets Europe S.L (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-021882-57
Record Dates: First submitted 2012-05-03; First posted 2012-05-10 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Tooth Extraction
Keywords: TT-173; Topical Hemostatics; Hemostasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- TT-173 (Experimental): TT-173
  Interventions: Drug: TT-173

INTERVENTIONS:
Drug: Placebo — It is applied directly to the bleeding site after tooth extraction
  Arms: Placebo
Drug: TT-173 — It is applied directly to the bleeding site after tooth extraction
  Arms: TT-173

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and efficacy of TT-173 in healthy volunteers after tooth extraction.

DETAILED DESCRIPTION:
As the TT-113 has been cleared for use as a topical hemostatic agent, the proposed study will further investigate the safety, tolerability and efficacy of TT-113 in healthy volunteers after tooth extraction.

ELIGIBILITY:
Inclusion Criteria:

* Subjects to be undertaken for the simple extraction of at least one tooth (incisor, canine, premolar, molar different of third molar) that cause bloody wound, located in the upper or inferior maxillary area of the mouth either
* Subjects who are able and willing to provide written and signed informed consent
* All subjects willing to use a medically accepted form of contraception from the time of consent to completion of all follow-up study visits. Negative pregnancy test result in the screening visit.

Exclusion Criteria:

* Subjects with personal and family history that could affect correct hemostasis
* Subjects with any clinically-significant coagulation disorder including including deficiencies in any of coagulation factors, thrombocytopenia and vascular purpura
* Subject with hipersensivity of TT-173 of any of its components or has a known allergy.
* Subjects who are unable to adequately follow or understand the instructions and requirements of the study.
* Subjects that are not fully free to give informed consent, or any other obstacle in the opinion of investigator support the conclusion that the subject is not fully reasoned.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 4 months

SECONDARY OUTCOMES:
Cmax, Tmax, AUC and bioavailability | 48 h
Determine the presence of coagulation disorders | 4 months
  Blood platelets, Prothrombin time, Fibrinogen, Thrombin time
Determine the immune responses to TT-173 | 4 months
  Antibody concentration
Time to hemostasis until cessation of bleeding | time 0 until cessation of bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Thrombotargets Europe SL, Castelldefels, Barcelona, Spain

REFERENCES:
- See also: Related Info — http://www.thrombotargets.com